CLINICAL TRIAL: NCT06487741
Title: Efficacy of a Home-based Stretching Program on Fibromyalgia Symptoms: a Randomised Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College of Northern Denmark (Other)
Collaborators: Bispebjerg Hospital (Other); University of Copenhagen (Other); Aalborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Fibromyalgia RCT
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2024-11

CONDITIONS: Fibromyalgia; Stretch; Adherence, Treatment
Keywords: Fibromyalgia; Stretching exercises; Home-based; Adherence
MeSH Terms: conditions — Fibromyalgia; Treatment Adherence and Compliance

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are blinded to the results of the pressure pain threshold measurements. Participants and the outcome assessor are blinded to the range of motion measurement results. The outcome assessor (MPS) is blinded to the outcome of the FIQ-R, SF-36 and IPAQ questionnaires.
  Blinding participants and the care provider (MPS) from delivering the intervention from treatment allocation is contrary to the nature of the investigated intervention and, therefore, is not considered feasible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group receives a home-based rehabilitation program consisting of six weeks of daily static stretching exercises (six minutes a day).
  Interventions: Other: Home-based stretching exercises
- Control (No Intervention): The control group receives usual care, and no change in treatment is made. Participants will be encouraged to maintain their daily routine but refrain from changing the current pharmacological treatment or initiating new physical exercise practices during the study.

INTERVENTIONS:
Other: Home-based stretching exercises — The intervention comprises six weeks of daily static stretching exercises (six minutes a day) in accordance with the recommendation of the American College of Sports Medicine. The intervention is self-administered and consists of two bouts of 30-second bilateral static stretches of the knee flexors, hip abductors, and shoulder elevators.
  Arms: Intervention

SUMMARY:
This randomised controlled trial will examine the clinical efficacy of a six-week, novel, home-based stretching programme compared to usual care on the effect of symptoms experienced by patients with fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* individuals diagnosed with fibromyalgia in accordance with the ACR 2016 diagnostic criteria.
* individuals diagnosed with chronic non-malignant pain or individuals diagnosed with chronic widespread pain (including fibromyalgia syndrome) are also included when they meet the ACR 2016 diagnostic criteria.

Exclusion Criteria:

* Non-controlled systemic disorders (such as hypertension, diabetes and coronary insufficiency),
* neurological conditions that impair alertness or comprehension, musculoskeletal conditions that could compromise assessments (such as nerve root compression or knee joint inflammation),
* relevant joint disorders (such as severe arthritis, arthroplasty of the hip or knee, and rheumatoid arthritis),
* recent changes in therapy for fibromyalgia (i.e., within four weeks of baseline).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Severity of symptoms | Measured at baseline
  The Revised Fibromyalgia Impact Questionnaire (FIQ-R) total score
Severity of symptoms | Measured following 6 weeks of intervention (primary endpoint)
  The Revised Fibromyalgia Impact Questionnaire (FIQ-R) total score
Severity of symptoms | Measured 6 months after the primary endpoint (secondary endpoint)
  The Revised Fibromyalgia Impact Questionnaire (FIQ-R) total score

SECONDARY OUTCOMES:
Health-Related Quality of life (HRQL) | Measured at baseline
  HRQL is assessed using the Danish version of the Short Form-36
Health-Related Quality of life (HRQL) | Measured following 6 weeks of intervention (primary endpoint)
  HRQL is assessed using the Danish version of the Short Form-36
Health-Related Quality of life (HRQL) | Measured 6 months after the primary endpoint (secondary endpoint)
  HRQL is assessed using the Danish version of the Short Form-36
Self-reported physical activity | Measured at baseline
  The International Physical Activity Questionnaire (IPAQ) short form
Self-reported physical activity | Measured following 6 weeks of intervention (primary endpoint)
  The International Physical Activity Questionnaire (IPAQ) short form
Self-reported physical activity | Measured 6 months after the primary endpoint (secondary endpoint)
  The International Physical Activity Questionnaire (IPAQ) short form
Range of motion | Measured at baseline
  Passive knee extension range of motion is assessed using the Biodex System 4 Pro isokinetic dynamometer
Range of motion | Measured following 6 weeks of intervention (primary endpoint)
  Passive knee extension range of motion is assessed using the Biodex System 4 Pro isokinetic dynamometer
Pain sensitivity | Measured at baseline
  Pain sensitivity expressed as pressure pain thresholds are assessed using a handheld electronic pressure algometer
Pain sensitivity | Measured following 6 weeks of intervention (primary endpoint)
  Pain sensitivity expressed as pressure pain thresholds are assessed using a handheld electronic pressure algometer

OTHER OUTCOMES:
Adherence | Measured following 6 weeks of intervention (primary endpoint)
  Adherence to the intervention is evaluated by the number of days stretching is performed using the self-reported data from the mHealth app.

CONTACTS AND LOCATIONS:
Overall Officials: Lise Eckardt, Pt. Msc, Study Director — Department of Physiotherapy, University College of Northern Denmark
Locations (1):
- University College of Northern Denmark, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Yes
The study protocol will be published open access. Data is made available upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: The study protocol will be published open access.
Access Criteria: Data is made available upon request.

REFERENCES:
- [Derived] Stove MP, Magnusson SP, Thomsen JL, Riis A. Efficacy of a home-based stretching programme on fibromyalgia symptoms: study protocol for a randomised controlled trial. Trials. 2025 Feb 27;26(1):74. doi: 10.1186/s13063-025-08776-z. PMID 40016827